CLINICAL TRIAL: NCT05312762
Title: An Open Label, Multicentre, Randomized Phase IV Clinical Trial to Evaluate the Safety and Efficacy of MaxioCel Compared With Aquacel Extra for the Management of Exuding Chronic Wounds
Brief Title: To Evaluate the Efficacy and Safety of MaxioCel Versus Aquacel Extra for the Management of Chronic Wounds
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Axio Biosolutions Pvt. Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABSPL/01/2021
Record Dates: First submitted 2022-03-18; First posted 2022-04-05 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Wound
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MaxioCel (Experimental): Microfiber wound dressing
  Interventions: Device: MaxioCel
- AquaCel Extra (Active Comparator): Hydrofiber dressing
  Interventions: Device: AquaCel Extra

INTERVENTIONS:
Device: MaxioCel — Microfiber wound dressing
  Other Names: Chitosan Wound Dressing
  Arms: MaxioCel
Device: AquaCel Extra — Hydrofiber dressing
  Arms: AquaCel Extra

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of MaxioCel vs Aquacel Extra in the management of exuding ulcers/wounds over a period of 4 weeks

DETAILED DESCRIPTION:
The current study intends to compare the efficacy of the chitosan wound dressing (MaxioCel) with another marketed dressing (Aquacel Extra). MaxioCel is made up of chitosan and Aquacel Extra with carboxymethyl cellulose. Both are polymeric dressings.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years old or above (till 80 years)
* Patients who are willing to sign the written informed consent
* Clinically diagnosed with an unhealed or non-healing diabetic foot ulcer / venous ulcer / arterial ulcer / other ulcers / wounds, etc.
* Wound duration between 1 to 24 months
* A target wound area between 1 cm2 and 50 cm2
* Exuding wounds / ulcers

Exclusion Criteria:

* Known allergy/hypersensitivity to the dressing
* Pregnant women
* Underlying or diagnosed with serious diseases or deemed unsuitable for this clinical study by the study's clinician
* Dry wounds
* Being treated with a high dose of steroids or immunosuppressant therapy or systemic antibiotics
* Presenting a progressive neoplastic lesion treated with radiotherapy or chemotherapy
* Patients who had Deep Vein Thrombosis in the previous 3 months
* Ulcers with clinical signs of infection or erysipelas of the lower limb or biofilm
* Subjects included in clinical study at present or during the past 30 days
* Clinical suspicion of osteomyelitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2022-04-27 (Actual); Primary Completion 2023-12-11 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Wound Area Measurement | Week 1, Week 2, Week 3, Week 4
  Wound area (cm2) to be recorded at baseline and weekly visits to assess % change in wound area.

SECONDARY OUTCOMES:
Pain Management | Week 1, Week 2, Week 3, Week 4
  Changes in pain using Numeric Rating Scale (0-10). 0 means no pain, 10 means severe pain/worst possible pain
Exudate Management | Week 1, Week 2, Week 3, Week 4
  Change in Exudate levels will be evaluated. Exudate levels will be evaluated as per below categories:
  None, Scant, Small, Moderate, Large
Changes in Epithilizing / Granulating Tissues | Week 1, Week 2, Week 3, Week 4
  measured by % change in Epithelizing and granulating tissues
Bates Janesen Wound Assessment Score | Week 1, Week 2, Week 3, Week 4
  The status of wound as per 13 items mentioned in the Bates-Jensen Wound Assessment Tool will be evaluated. Higher the total score, the more severe the wound status.Minimum score - 13 ; Maximum score - 65
Scar Management | Week 4
  Vancouver Scar Scale will be used at the final visit to evaluate the scar formation at wound site. Minimum score - 0; Maximum score - 13
Clinician opinion related to dressing | Week 4
  Dressing usability / use of dressing will be evaluated via questionnaire. The options for rating will be Excellent, Good, Fair, Poor. For few questions, options will be Yes or No
Patient opinion related to dressing | Week 4
  Patients comfort levels with use of dressing will be evaluated via questionnaire. The options for rating will be Excellent, Good, Fair, Poor. For few questions, options will be Yes or No

CONTACTS AND LOCATIONS:
Overall Officials: Shailee Mehta, MSc, Study Chair — Axio Biosolutions Pvt. Ltd.
Locations (5):
- India (5):
  - Hycare Super Speciality Hospital, Chennai, Tamil Nadu
  - Saveetha Medical College Hospital, Chennai, Tamil Nadu
  - Vijaya hospitals, Chennai
  - Kamineni Hospitals Pvt Ltd, Hyderabad
  - Yalamanchi hospital and research center vijayawada, Vijayawada

IPD SHARING:
Plan to Share IPD: No